CLINICAL TRIAL: NCT05255198
Title: Anterior Minimal Invasive Surgery Versus Antero-lateral Approach in Hip Joint Hemiarthroplasty
Status: Completed | Type: Observational
Sponsor: Rehabilitation Hospital Tobelbad (Other)
Responsible Party: Principal Investigator, Renate Krassnig MD PhD, Consultant, Rehabilitation Hospital Tobelbad
Other Study IDs: HHAP$1
Record Dates: First submitted 2021-08-30; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Arthroplasty; Clinical Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterolateral approach
  Interventions: Procedure: Anterior versus lateral approach to hip joint
- Direct anterior approach
  Interventions: Procedure: Anterior versus lateral approach to hip joint

INTERVENTIONS:
Procedure: Anterior versus lateral approach to hip joint

SUMMARY:
Comparison between two minimally invasive approaches to the hip joint.

DETAILED DESCRIPTION:
Following parameters were compared: modified Barthel-Index, pain, complications, developing of heterotopic ossification.

ELIGIBILITY:
Exclusion Criteria:

Exclusion criteria represented acute local or systemic infection, open or pathological fractures, concomitant injuries of the ipsi- or contralateral leg and rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients, presenting with indication for bipolar hemiarthroplasty of the hip joint due to Garden III and IV fractures, who had given their written informed consent, were enrolled in the study. Exclusion
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | one year after surgery
  Pain score

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05255198/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05255198/ICF_001.pdf